CLINICAL TRIAL: NCT00114855
Title: A Single-Centre, Randomised Double-Blind Placebo-Controlled Study to Measure the Effect of Hypocol® on Lipids in Subjects With Mild Hypercholesterolemia and Mildly Elevated Blood Glucose
Brief Title: The Effect of Hypocol® on Lipids in Subjects With Mild Hypercholesterolemia and Mildly Elevated Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Pharmalogica (Industry); Wearnes Biotech @ Medicals (Unknown); Beijing Peking University WBL Biotech Co., Ltd. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HYPOCOL protocol 15.12.2004; S-04329 (REK Sør); 11850 (NSD); 05/896 TSP (ShDir); 200303963-3 (SLV)
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-02

CONDITIONS: Hyperlipidemia; Glucose Metabolism Disorders
Keywords: Hypocol; Red yeast rice; Patients with mild Type IIa, Type IIb or IV hyperlipidaemia (LDL-cholesterol >3.0 mmol/L< 6.0 mmol/L.; Mildly elevated blood glucose
MeSH Terms: conditions — Hyperlipidemias; Glucose Metabolism Disorders

INTERVENTIONS:
Drug: HYPOCOL®

SUMMARY:
The purpose of this study is to determine to what degree Hypocol® (Red Yeast Rice) may lower low density lipoprotein (LDL)-cholesterol in a European population. The effect of Red Yeast Rice on fasting blood glucose and inflammatory markers will also be investigated.

DETAILED DESCRIPTION:
Clinical end-point trials have demonstrated that lowering cholesterol levels with statins reduces the incidence of cardiovascular events and mortality. Subgroup analyses of the large clinical studies, the West of Scotland Coronary Prevention (WOSCOP) and Cholesterol and Recurrent Events (CARE), have suggested that the beneficial effects of statins may extend to mechanisms beyond cholesterol reduction. A variety of mechanisms accounting for these effects have been suggested. Among these, the anti-inflammatory activity is particularly attractive because inflammation is considered an early step in the development of atherosclerosis. Thus, statin therapy has been shown to lower high-sensitivity C-reactive protein (CRP), a plasma marker of inflammation, in hypercholesterolemic patients. Furthermore, statins may possess anti-inflammatory properties by their ability to reduce the number of inflammatory cells in atherosclerotic plaques. Red Yeast Rice contains Lovastatin and lowers LDL-cholesterol. However, it is not known to what degree Red Yeast Rice may lower LDL-cholesterol in a European population. Some reports have suggested an effect of Red Yeast Rice on fasting blood glucose by an unknown mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to enrolment (any study-specific procedures or investigations).
* Male or female aged between 18 and 75 years.
* Patients with mild Type IIa, Type IIb or IV hyperlipidaemia (LDL-cholesterol >3.0 mmol/L< 6.0 mmol/L)
* Fasting serum TG level < 4.5 mmol/L
* Mildly elevated blood glucose defined as at least one of three of the following criteria

  * HbA1c% >5.5% < 7.5%;
  * Fasting glucose > 5.5 mmol/L;
  * Type 2 diabetes mellitus on stable oral antihyperglycemic treatment for more than 8 weeks and HbA1c% < 7.5% at the time for inclusion.
* If female, be of non-childbearing potential, i.e., post-menopausal (defined as >12 months since last menstrual period) or surgically sterilised, or using adequate barrier contraception if of childbearing potential.

Exclusion Criteria:

* Currently taking lipid-lowering medication and are not able to complete the 4-week wash-out prior to the start of the dietary run-in period.
* History of active malignant disease the last 5 years (excluding treated basal cell carcinoma).
* History of infection with human immunodeficiency virus (HIV) or hepatitis B or C.
* History of alcohol and/or drug abuse.
* Have uncontrolled hypertension (diastolic blood pressure >100 mmHg). Patients who are taking antihypertensive medication will not be excluded provided they are maintained at a stable dose for 3 months prior to screening and the stable dose is maintained throughout the study.
* Have uncontrolled thyroid disease (thyroid dysfunction controlled for at least 6 months prior to screening is permitted).
* Known homozygous familial hypercholesterolaemia or known Type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia).
* Patients with active liver disease or hepatic dysfunction as defined by elevations in liver enzymes [alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyltransferase (GGT) and alkaline phosphatase (ALP)] or total bilirubin >2 x the upper limit of normal (ULN) at any time between Visit 1 (Week -4) and Visit 3 (Week -1).
* Patients with a serum creatinine >180 µmol/L at any time between Visit 1 (Week -4) and Visit 3 (Week -1)
* Patients who have serious or unstable medical or psychological conditions which, in the opinion of the investigator, would compromise the patient's safety or successful participation in the study.
* Patients who started hormone replacement therapy (HRT) less than 6 months prior to screening.
* Currently taking other investigational drugs or have taken part in a clinical trial within the previous 30 days prior to screening.
* These drugs should not be given during the patient's participation in the study, and must be stopped 6 weeks before randomisation : lipid lowering drug other than study medication, Cyclosporine A, medical treatment against obesity (i.e., Orlistat, Sibutramine), oral anticoagulants. Special attention will be paid to the medications that could interfere with the lipid profile (i.e. oral corticosteroids, retinoids, thyroid hormones, thiazide derivative, diuretics, beta-blockers, and hormone replacement therapies). It is recommended not to modify these medications within 6 weeks prior to study start and during the course of the trial (unless this is medically required). All concomitant medications will be recorded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The effect of HypoCol on lipids in subjects with mild hypercholesterolemia.

SECONDARY OUTCOMES:
The effect of HypoCol on fasting glucose, glycosylated hemoglobin (HbA1c) and high sensitive CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Retterstøl, Dr. med, Principal Investigator — Oslo University Hospital
Locations (1):
- Lipidklinikken, Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Bogsrud MP, Ose L, Langslet G, Ottestad I, Strom EC, Hagve TA, Retterstol K. HypoCol (red yeast rice) lowers plasma cholesterol - a randomized placebo controlled study. Scand Cardiovasc J. 2010 Aug;44(4):197-200. doi: 10.3109/14017431003624123. PMID 20636227